CLINICAL TRIAL: NCT05110833
Title: Dose Responsiveness as a Measure of Clinical Effectiveness During Neuromonitored Spine Surgery
Acronym: IONM
Status: Enrolling by invitation | Type: Observational
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 1557758
Record Dates: First submitted 2021-09-09; First posted 2021-11-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Spinal Curvatures; Spinal Stenosis; Spondylitis; Spondylosis
Keywords: IONM
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Spinal Curvatures; Spinal Stenosis; Spondylitis; Spondylosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intraoperative Neuromonitoring (IONM) is a tool used by neurophysiologists during spine surgery to prevent irreversible damage to the spinal cord during procedures through a system of alerts. This study investigates the effectiveness of IONM in 300 participants receiving spine surgery. The goal of this study is to refine the alert criteria for procedures in which IONM is used.

DETAILED DESCRIPTION:
Intraoperative neurophysiological monitoring (IONM) measures neural function and integrity during surgical procedures. Through IONM, neurodiagnostic procedures can help determine whether any nerves have become compressed or if the brain or spinal cord has any reduced vascular flow, allowing the surgical team to take immediate and corrective actions to prevent a bad outcome. Essentially, IONM acts as an early warning system for surgeons to gain reliable insight into a patient's condition during surgery, adding a layer of safety to the measures already in place that monitor cardiac and respiratory function while a patient is anesthetized.

We propose an observational research study to enhance the evidence-base for IONM. A novel prospective neuromonitoring database will be implemented. In addition to the usual contingency data to assess prediction accuracy, other measures will be examined:

1. A "dose effect of injury" assessment. Three categories of injury will be recorded by physicians: (a) No New Deficit; (b) New Minor Deficit; and (c) New Severe Deficit.
2. The outcome effect of intraoperative test frequency will be evaluated (infrequent vs average vs very frequent), leading to a "dose effect of neuromonitoring" assessment. Here we hypothesize that within our prospective sample, there is a relationship between the proportion of total new neurological deficits (New Minor Deficit + New Severe Deficit) and the frequency of IONM testing. More frequent testing is associated with fewer total new neurological deficits.
3. Patient reported outcomes will be evaluated longitudinally in conjunction with clinical outcomes data. Patient interviews will be conducted by a trained research assistant aided by department technologists. Patient-reported neurological outcome assessments will be supplemented/confirmed by review of in- and outpatient surgical/neurophysiologist physician chart notes.

Data from this proposed observational study will allow real-life outcomes based improvement in the field of IONM.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18+ years old
* Patients must be undergoing cervical and/or thoracic spine surgical procedure at Abbott Northwestern Hospital in Minneapolis, MN

Exclusion Criteria:

* Patients who are non-English speakers
* Patients with ongoing psychiatric concerns are excluded
* Patients unwilling to be contacted for a 6-month follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anyone 18 or older of any sex undergoing cervical and/or thoracic spine surgical proceudre with intraoperative neuromonitoring at Abbott Northwestern Hospital in Minneapolis, MN
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Nature of changes in free-run smooth muscle EMG under varying surgical and anesthetic conditions | 1 day
  Free-run smooth muscle EMG will be monitored continuously throughout the duration of surgery. Any changes in the EMG, as indicated by fluctuation in amplitude and/or frequency, will be recorded.
Nature of changes in free-run smooth muscle EMG resulting from the inadvertent effect of intraoperative monitoring stimulation and recording. | 1 day
  Smooth muscle EMG in response to stimulations and recordings will be monitored. Any changes in the EMG, as indicated by fluctuation in amplitude and/or frequency, will be recorded.
The believable and repeatable smooth muscle EMG response, if any, measured by amplitude and frequency after deliberate spinal/extra-spinal neural stimulations. | 1 day

SECONDARY OUTCOMES:
Short Form (36) Health Survey | 1 year
  A self-report survey of patient health

CONTACTS AND LOCATIONS:
Overall Officials: Stanley A Skinner, MD, Principal Investigator — Allina Health
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No